CLINICAL TRIAL: NCT05510388
Title: High-flow Nasal Cannula Oxygenation Reduces the Incidence of Hypoxia During Gastroscopy or Colonoscopy Sedated With Propofol in High-risk Patients: a Multi Central Randomized Controlled Study
Brief Title: HFNO Reduces Hypoxia During Sedated Gastroscopy or Colonoscopy in High Risk Patients
Acronym: HRISK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2022-116-B
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer; Intestinal Cancer; Intestine Adenoma; Gastritis
Keywords: Gastroscopy; High-flow nasal oxygenation; Hypoxia; High-risk; Colonoscopy
MeSH Terms: conditions — Stomach Neoplasms; Intestinal Neoplasms; Gastritis; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula oxygenation group (Experimental)
  Interventions: Device: High-flow nasal cannula oxygenation
- Regular nasal cannula oxygenation group (Active Comparator)
  Interventions: Device: Regular nasal cannula oxygenation

INTERVENTIONS:
Device: High-flow nasal cannula oxygenation — The patients receive oxygen flow of 6L/min for preoxygenation with an high-flow canular oxygenation device before losing of conscious. Then, the oxygen flow is adjusted to 60L/min with the oxygen concentration of 100% and the temperature of 37℃ until the end of procedure.
  Arms: High-flow nasal cannula oxygenation group
Device: Regular nasal cannula oxygenation — The patients receive an oxygen flow of 6L/min for preoxygenation with a disposal regular nasal cannula until the end of procedure.
  Arms: Regular nasal cannula oxygenation group

SUMMARY:
The objective of this study is to observe the preventive effects of high flow nasal oxygenation on the incidence of hypoxia during gastroscopy or colonoscopy sedated with propofol in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 to 80, both sexes
2. Patients receiving selective gastroscopy or colonoscopy or gastroscopy and colonoscopy procedure
3. ASA Ⅲ~Ⅳ
4. 18 kg/m2<BMI<28kg/m2
5. The anticipated operation time of the procedure shall be less than 30min.
6. Patients should clearly understand and voluntarily participate in the study, with signed informed consent.

Exclusion Criteria:

1. Patients with nasal congestion, epistaxis, recent nasal trauma, recent nasal surgery, increased intracranial pressure and skull fracture, etc. who can not tolerate high-flow nasal cannula.
2. Patients diagnosed POCD
3. Patients clearly identified difficult airway
4. Patients with mechanical ventilation
5. Patients with acute respiratory infection and asthma
6. Patients with acute upper gastrointestinal hemorrhage accompanied by shock, severe anemia, gastrointestinal obstruction accompanied by retention of gastric contents
7. Patients with aortic stenosis and carotid stenosis
8. Patients allergic to sedatives such as propofol
9. Patients without civil capacity such as cognitive dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Hypoxia refers to 75%≤SpO2<90%,<60S

SECONDARY OUTCOMES:
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Severe hypoxia refers to SpO2<75% lasting for any time, or 75%≤SpO2<90%, ≥60s
The incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Subclinical respiratory depression refers to 90%≤ SpO2<95%
Other adverse events evaluated by the tool of World SIVA | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
Complications related to high-flow nasal cannula | Patients will be followed for the duration of hospital stay, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Hospital Affiliated to Chongqing Medical University, Chongqing, Chongqing Municipality
  - Henan Provincial people's hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No